CLINICAL TRIAL: NCT04926220
Title: Estimation of Cardiac Output in the Operating Room by Pulse Wave Analysis and Esophageal Doppler Blood Velocity: Comparison of the Two Methods
Brief Title: Dynamic Estimation of Cardiac Output in the Operating Room
Acronym: TRIPLEFLOW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210311; 2021-A00088-33 (Other: IDRCB)
Record Dates: First submitted 2021-06-07; First posted 2021-06-15 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-06

CONDITIONS: Interventional Radiology; Surgery; General Anesthesia; Organ Failure; Intensive Care; Hemodynamic Instability; Blood Pressure; Cardiac Output
Keywords: Cardiac output monitoring; Pulse contour analysis; Vasopressors; Fluid challenge; Trans-esophageal doppler; Pressure recording analytical method; Long time interval analysis
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing general anesthesia and benefiting from intraoperative hemodynamic optimization: Patients undergoing general anesthesia and benefiting from intraoperative hemodynamic optimization, including routine monitoring of blood pressure and measurement of cardiac output by trans-esophageal Doppler.
  Interventions: Device: Trans-esophageal Doppler monitoring; Device: MostCareUP Haemodynamic Monitor; Device: Argos Cardiac Output (CO) Monitor

INTERVENTIONS:
Device: Trans-esophageal Doppler monitoring — Trans-esophageal Doppler monitoring (CARDIOQ-ODM; Deltex Medical, Chichester, UK) for monitoring of cardiac output
Device: MostCareUP Haemodynamic Monitor — MostCareUp (Vytech, Padova, Italy) waveform analysis cardiac output monitor
Device: Argos Cardiac Output (CO) Monitor — Argos monitor (Retia Medical, Valhalla, NY, USA) for cardiac output monitoring

SUMMARY:
During major surgery, it is recommended to monitor invasive arterial blood pressure and cardiac output (CO) during hemodynamic interventions (fluid challenge or vasopressors). Esophageal Doppler is currently considered as the reference method for monitoring cardiac output in the operating room. The PRAM method (pressure recording analytical method) with the MostCareUp monitor (Vytech, Padova, Italy) and the LTIA method (long time interval analysis) allow cardiac output estimation derived from non-calibrated arterial pressure waveform analysis. Few studies have looked at relative changes in cardiac output during hemodynamic intervention with these two methods. The aim of this study is to compare the relative changes in cardiac output during hemodynamic interventions as measured using PRAM and LTIA methods, compared to esophageal Doppler.

DETAILED DESCRIPTION:
Hemodynamic optimization is a major issue in the perioperative and intensive care settings. The titration of fluid in the operating room and in intensive care guided by the variations of the stroke volume (SV) and therefore of the cardiac output (CO) improves morbimortality. Esophageal Doppler is currently considered as the reference method for monitoring cardiac output in the operating room. However, when its use is not possible, there are devices that allow continuous estimation of cardiac output from the pulse wave contour (i.e. an invasive blood pressure signal). The PRAM method (pressure recording analytical method) with the MostCareUp monitor (Vytech, Padova, Italy) and the LTIA method (long time interval analysis) using an analog-to-digital converter connected to the patient's scope seem to be promising pulse wave analysis techniques. The majority of studies investigating these devices have focused on cardiac output values from a purely static perspective. Few studies have looked at changes in cardiac output during hemodynamic intervention (fluid challenge or use of vasopressors). However, in daily clinical practice, it is the dynamic information on CO that informs doctors on the effectiveness of therapeutic challenges. Thus, our hypothesis is to compare the variations in cardiac output estimated by PRAM et LTIA methods with those obtained using esophageal Doppler, during surgical procedures under general anesthesia.

The main goal of this study is to compare the relative changes in cardiac output obtained during hemodynamic interventions (fluid challenge or vasopressors) using PRAM and LTIA versus esophageal doppler. Parameters measured for the primary objective: 1. Continuous measurement and recording of the invasive blood pressure signal 2. Continuous and simultaneous measurement of cardiac output by MostCareUp (Vytech, Padova, Italy) and esophageal doppler. 3. Estimation of cardiac output from the arterial pressure signal by means of a digital analog converter using the LTIA algorithm connected to the patient's scope. For all patients, data from the cardiac output monitors are recorded throughout the procedure and the resuscitation stay. The secondary objective is to study the hemodynamic parameters of ventriculoarterial coupling calculated by the PRAM method and measured by esophageal doppler, other than CO and SV during therapeutic challenges. Parameters measured for the secondary objective: Global Afterload Angle (GALA), the value of the dicrote wave, dP/dtmax (myocardial contractility index), cardiac efficiency (CCE), arterial elastance, the total impedance of the system (Ztot).

Experimental design: this is a single-center, observational prospective study The study concerns adult patients benefiting from intraoperative hemodynamic optimization under general anesthesia, including routine monitoring of blood pressure and measurement of cardiac output by esophageal Doppler.

This study is "non-interventional" on adult patients undergoing interventional radiology, surgery under general anesthesia, or admitted to the ICU for postoperative organ failure. All measurements are obtained from standard monitoring including blood pressure and cardiac output measurement by transesophageal Doppler. Monitoring includes continuous electrocardiogram, SpO2, ventilatory parameters and depth of anesthesia by Bispectral Index. During the anaesthesia consultation, the patients will be given a letter of information on the objectives and the course of the study. Their non-opposition to participating in this study will be collected at the latest during the pre-anesthetic visit, the day before the operation. The protocol starts on the day of the operation. For all patients, the procedures will be performed under general anesthesia with an intravenous anesthesia protocol with a concentration objective (Orchestra® Base Primea - Fresenius Kabi France). The protocol does not interact with the care procedure. On the day of the procedure, the MostCareUp (Vytech, Padova, Italy) will be connected in series with the pressure head already in place. The blood pressure signals will be continuously recorded to allow estimation of the cardiac output by the LTIA method using an analog-to-digital converter. This calculation is made from the signal that has been transmitted to the multiparametric scope monitor and is therefore not directly connected to the patient. The acquisition of the analog signal is done via USB2.0 thanks to a Video Capture Card equipped with a converter. The software recalculates with its algorithm an estimation of the cardiac output from the data. The clinician in charge in the operating room will use only the hemodynamic data from the esophageal Doppler to guide his therapeutic strategy. Synchronization of the 2 devices. Recording of events during therapeutic tests if there is an indication for treatment. Usual protocol of the therapeutic challenges service: Patient receiving intraoperative vascular filling titration to optimize cardiac output (maximize SV/CO), patient with persistent arterial hypotension (MAP < 65 mmHg or < 80% of baseline) during the procedure despite adequate depth of anesthesia (BIS 40-50) and optimized cardiac output motivating vasopressor injection. For all patients, data from the 2 cardiac output monitors and hemodynamics will be collected during and after the therapeutic tests. Under no circumstances will a decision on therapeutic strategy be made based on PRAM or LTIA data. No additional complementary examination will be performed. The physician in charge of the study collecting the data does not intervene at any time in the management of the patient. The implementation of this type of intraoperative monitoring does not prolong the duration of anesthesia.

The measure of agreement the investigators will use is the intra-class correlation coefficient. To compare 3 measurement modalities, assuming that the intraclass correlation coefficient for the measurement of VES variations will be 0.85 with a confidence interval with width of 0.1 and a first-species risk of 0.05, 84 patients must be included. It is expected that the signals of 10% of the included patients will be of insufficient quality for their exploitation. Therefore, the calculated sample size is 92 patients.

Results will be expressed as mean (standard deviation) or median (interquartile range) depending on the normality of the data distribution. A Bland-Altman analysis for repeated measures will be used to evaluate the agreement between the cardiac output measured by esophageal Doppler and the cardiac output estimated by the two pulse wave monitors. It will be associated with a calculation of the bias and its 95% confidence interval, the upper/lower limits of agreement and their 95% confidence intervals, and the percentage error. A percentage of error less than or equal to 30% indicates the agreement of the technique with the reference method. The agreement of cardiac output variations measured by esophageal Doppler and pulse wave analysis will be evaluated by a Bland-Altman analysis. The percentage of agreement will be evaluated using a four-quadrant plot. Acceptable agreement is defined as greater than 90%. The analyses will be repeated in the filler and vasopressor subgroups. The ability of pulse wave monitors to detect responders to filling will be assessed and compared with esophageal doppler. Subjects will be defined as responders to volume expansion when the filling test increases the ESV by more than 10%.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (≥ 18 years )
* Eligible for an interventional radiology procedure or surgery under general anesthesia
* Monitoring of invasive blood pressure and cardiac output by trans-esophageal Doppler.
* Patients informed and having expressed their non-opposition to participation in this research

Exclusion Criteria:

* Patients under 18 years old
* Atrial fibrillation
* Contraindication to trans-esophageal doppler
* Patient opposed to protocol participation
* Pregnant woman
* Patient under judicial protection
* Patient without affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients eligible for an interventional radiology procedure, surgery under general anesthesia, or admitted to intensive care unit for postoperative organ failure, benefiting from intraoperative and postoperative hemodynamic optimization in intensive care including routine blood pressure monitoring and measurement of cardiac output by esophageal Doppler.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac output using the trans-esophageal Doppler technique | Duration of the surgery (maximum 1 day)
  Measure of cardiac output with trans-esophageal doppler (CARDIOQ-ODM; Deltex Medical, Chichester, UK) in L/min (COTOD)
Cardiac output using the MostCareUp monitor | Duration of the surgery (maximum 1 day)
  Measure of cardiac output with MostCareUp (Vytech, Padova, Italy) in L/min (COPRAM)
Cardiac output using the Argos monitor | Duration of the surgery (maximum 1 day)
  Measure of cardiac output with Argos monitor (Retia Medical, Valhalla, NY, USA) in L/min (COLTIA)

SECONDARY OUTCOMES:
Measure of the value of the dicrote wave with MostCareUp monitor | Duration of the surgery (maximum 1 day)
  The value of the dicrote wave will be recorded with the MostCareUp monitor (Vytech, Padova, Italy) during the whole procedure
Measure of dP/dtmax (myocardial contractility index) with MostCareUp monitor | Duration of the surgery (maximum 1 day)
  The dP/dtmax (myocardial contractility index) will be recorded with the MostCareUp monitor (Vytech, Padova, Italy) during the whole procedure
Measure of the cardiac efficiency (CCE) with MostCareUp monitor | Duration of the surgery (maximum 1 day)
  The cardiac efficiency (CCE) will be recorded with the MostCareUp monitor (Vytech, Padova, Italy) during the whole procedure
Measure of arterial elastance with MostCareUp monitor | Duration of the surgery (maximum 1 day)
  The arterial elastance will be recorded with the MostCareUp monitor (Vytech, Padova, Italy) during the whole procedure
Measure of the total impedance of the system (Ztot) with MostCareUp monitor | Duration of the surgery (maximum 1 day)
  The total impedance of the system (Ztot) will be recorded with the MostCareUp monitor (Vytech, Padova, Italy) during the whole procedure
Measure of the Global Afterload Angle (GALA) using the trans-esophageal Doppler technique | Duration of the surgery (maximum 1 day)
  The Global Afterload Angle (GALA) will be recorded with trans-esophageal Doppler (CARDIOQ-ODM; Deltex Medical, Chichester, UK) during the whole procedure
Measure of arterial elastance using the trans-esophageal Doppler technique | Duration of the surgery (maximum 1 day)
  The the arterial elastance will be recorded with trans-esophageal Doppler (CARDIOQ-ODM; Deltex Medical, Chichester, UK) during the whole procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alex HONG, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care, Paris, France

IPD SHARING:
Plan to Share IPD: No